CLINICAL TRIAL: NCT00456508
Title: Open-label Patient Continuation of DX-88 (Ecallantide) for Acute Hereditary Angioedema Attacks
Brief Title: Safety and Efficacy Study of Repeated Doses of DX-88 (Ecallantide) to Treat Attacks of Hereditary Angioedema (HAE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DX-88/19
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2012-12-28 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — ecallantide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DX-88 (ecallantide) (Experimental): DX-88 (ecallantide) Patients were treated with DX-88 (ecallantide) when they experienced an HAE attack. 30 mg dose of ecallantide given via 3 SC injections; a second 30 mg dose can be administered if needed. Patients were to be assessed until 4 hrs post-dose. Patients were asked to return for 3 follow-up visits: 7 days, 28 days and 90 days post-dose.
  Interventions: Drug: ecallantide

INTERVENTIONS:
Drug: ecallantide — solution for SC injection, one 30 mg dose per HAE attack
  Other Names: DX-88

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of repeated doses of ecallantide in the treatment of acute attacks of hereditary angioedema and to allow HAE patients continued access to ecallantide. In addition, patients enrolled in DX-88/20 (EDEMA4) trial will be followed up and treated for subsequent attacks in this trial.

DETAILED DESCRIPTION:
This is an open label trial.

The study is designed to assess the efficacy and safety of 30 mg subcutaneous ecallantide in the treatment of acute attacks of hereditary angioedema. This study is designed to provide efficacy and safety data on repeated use of ecallantide. These data are intended to support the marketing authorization of ecallantide in the treatment of acute attacks of hereditary angioedema. Efficacy and safety of ecallantide will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* 10 years of age or older
* Documented diagnosis of HAE (Type I or II)
* Willing and able to give informed consent
* Acute HAE attack at time of presentation

Exclusion Criteria:

* Receipt of an investigational drug or device, within 30 days prior to study treatment, other than DX-88 (ecallantide)
* Pregnancy or breastfeeding
* Receipt of non-investigational C1-INH or DX-88 within 72 hours of treatment
* Patients eligible for current, ongoing clinical trial in which DX 88 (ecallantide) is offered

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2010-06-01 (Actual); Study Completion 2010-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (41):
- United States (39):
  - Aaron Davis, Scottsdale, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Little Rock Allergy & Asthma Clinic, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Pacific Coast Allergy, Crescent City, California
  - Jacob Offenberger, Granada Hills, California
  - UCLA David Geffen School of Medicine, Department of Medicine, Los Angeles, California
  - Asthma and Allergy Associates, P.C., Colorado Springs, Colorado
  - Christiana Hospital, Christiana Care Health Services, Newark, Delaware
  - Georgetown University Medical Center, Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami, General Clinical Research Center, Miami, Florida
  - University of South Florida, Asthma, Allergy and Immunology Clinical Research Unit, Tampa, Florida
  - Roberson Allergy and Asthma, West Palm Beach, Florida
  - Family Allergy & Asthma Center, PC, Atlanta, Georgia
  - Allergy Center of Brookstone, Columbus, Georgia
  - University Consultants in Allergy and Immunology, Chicago, Illinois
  - Muncie Allergy Center, Muncie, Indiana
  - Kansas City Allergy & Asthma, Overland Park, Kansas
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Asthma and Allergy Institutes of Michigan, Clinton Township, Michigan
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - Nevada Access to Research and Education Society, Las Vegas, Nevada
  - University of Nevada School of Medicine, Reno, Nevada
  - UMDNJ- New Jersey Medical School, Newark, New Jersey
  - Allergy Partners of Albuquerque, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - University of Cincinnati, Division of Internal Medicine, Cincinnati, Ohio
  - Optimed Research, LLC, Columbus, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Asthma Allergy and Pulmonary Associates, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Highlands Allergy and Asthma Center, PC, Bristol, Tennessee
  - The Paull Allergy and Asthma Clinic, P.A, Bryan, Texas
  - AARA Research Center, Dallas, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Puget Sound Allergy, Asthma, & Immunology, Tacoma, Washington
- Allergy and Asthma Research Centre, Ottawa, Ontario, Canada
- Jordan University Hospital, Amman, Jordan

REFERENCES:
- [Derived] Rubinstein E, Stolz LE, Sheffer AL, Stevens C, Bousvaros A. Abdominal attacks and treatment in hereditary angioedema with C1-inhibitor deficiency. BMC Gastroenterol. 2014 Apr 9;14:71. doi: 10.1186/1471-230X-14-71. PMID 24712435
- [Derived] MacGinnitie AJ, Davis-Lorton M, Stolz LE, Tachdjian R. Use of ecallantide in pediatric hereditary angioedema. Pediatrics. 2013 Aug;132(2):e490-7. doi: 10.1542/peds.2013-0646. Epub 2013 Jul 22. PMID 23878046
- [Derived] Sheffer AL, MacGinnitie AJ, Campion M, Stolz LE, Pullman WE. Outcomes after ecallantide treatment of laryngeal hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2013 Mar;110(3):184-188.e2. doi: 10.1016/j.anai.2012.12.007. Epub 2013 Jan 5. PMID 23548529
- [Derived] Li HH, Campion M, Craig TJ, Soteres DF, Riedl M, Lumry WR, MacGinnitie AJ, Shea EP, Bernstein JA. Analysis of hereditary angioedema attacks requiring a second dose of ecallantide. Ann Allergy Asthma Immunol. 2013 Mar;110(3):168-72. doi: 10.1016/j.anai.2012.12.004. Epub 2013 Jan 8. PMID 23548526

RESULTS

PARTICIPANT FLOW:
Groups:
- DX-88 (Ecallantide): Patients were treated with DX-88 (ecallantide) when they experienced an HAE attack. 30 mg dose of ecallantide given via 3 SC injections; a second 30 mg dose can be administered if needed. Patients were to be assessed until 4 hrs post-dose. Patients were asked to return for 3 follow-up visits: 7 days, 28 days and 90 days post-dose.
Period: Overall Study
Arm/Group | DX-88 (Ecallantide)
Started | 147
Completed | 147
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: DX-88 (ecallantide)
Arm/Group | Treatment
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 98
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 141
  Canada | 1
  Jordan | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Symptom Complex Severity (MSCS) Score at 4 Hrs Post Dosing
Description: Mean Symptom Complex Severity (MSCS) score is a validated point-in-time measure of symptom severity. At baseline and 4 hrs, patients rated the severity on a categorical scale (0=normal, 1=mild, 2=moderate, 3=severe) for symptoms at each affected anatomical location. Ratings were averaged to obtain the MSCS score. A decrease in MSCS score reflected an improvement in symptoms; clinically meaningful improvement was indicated by a reduction in the score of 0.30 or more.
Time Frame: 4 hrs post dose after every episode
Population: All efficacy analyses were to be based on the safety population (all treated patients). Only those patients with non-missing severity and response assessment were included in the change in MSCS score.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DX-88 (Ecallantide)
Number analyzed (Participants) | 138
scores on a scale
  change in MSCS at 4 hrs episode 1 (n=138) | -1.04 (0.773)
  change in MSCS at 4 hrs episode 2 (n=98) | -1.06 (0.731)
  change in MSCS at 4 hrs episode 3 (n=73) | -1.07 (0.801)
  change in MSCS at 4 hrs episode 4 (n=52) | -1.15 (0.791)
  change in MSCS at 4 hrs episode 5 (n=38) | -1.16 (0.746)
  change in MSCS at 4 hrs episode 6 (n=32) | -1.07 (0.806)
  change in MSCS at 4 hrs episode 7 (n=25) | -1.24 (0.797)
  change in MSCS at 4 hrs episode 8 (n=22) | -1.31 (0.667)
  change in MSCS at 4 hrs episode 9 (n=22) | -1.20 (0.764)
  change in MSCS at 4 hrs episode 10 (n=16) | -1.27 (1.027)
  change in MSCS at 4 hrs episode 11 (n=16) | -1.22 (0.643)
  change in MSCS at 4 hrs episode 12 (n=12) | -1.36 (0.677)
  change in MSCS at 4 hrs episode 13 (n=12) | -1.10 (0.657)

2. Secondary Outcome: Treatment Outcome Score (TOS) at 4 Hrs Post Dosing, Based on the Patient Assessment of Baseline Severity of Symptoms
Description: The Treatment Outcome Score (TOS)is a validated measure of response to therapy. Response assessment for each symptom complex (internal head/neck, stomach/GI, genital/buttocks, external head/neck or cutaneous) was to be weighted based on the severity of symptom complexes at baseline. Severity assessment at baseline was rated on a categorical scale (1=mild, 2=moderate, 3=severe) for symptoms at each affected symptom complex. Response assessment of each symptom complex post-dosing relative to baseline used a scale (100=significant improvement, 50=improvement, 0=same). The weighted values were used to calculate the composite TOS. A TOS greater than 0 denotes an improvement in symptoms compared with baseline severity.
Time Frame: 4 hrs post dose after every episode
Population: All efficacy analyses were to be based on the safety population (all treated patients). Only those patients with non-missing severity and response assessment were included in the change in TOS score.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DX-88 (Ecallantide)
Number analyzed (Participants) | 140
scores on a scale
  TOS at 4 hrs for episode 1 (n=140) | 69.80 (35.378)
  TOS at 4 hrs for episode 2 (n=98) | 70.05 (40.639)
  TOS at 4 hrs for episode 3 (n=73) | 63.08 (42.840)
  TOS at 4 hrs for episode 4 (n=52) | 62.65 (42.802)
  TOS at 4 hrs for episode 5 (n=39) | 65.13 (34.858)
  TOS at 4 hrs for episode 6 (n=32) | 60.42 (40.866)
  TOS at 4 hrs for episode 7 (n=25) | 56.20 (34.229)
  TOS at 4 hrs for episode 8 (n=22) | 79.77 (24.663)
  TOS at 4 hrs for episode 9 (n=22) | 71.06 (37.270)
  TOS at 4 hrs for episode 10 (n=16) | 76.30 (23.556)
  TOS at 4 hrs for episode 11 (n=16) | 60.94 (45.615)
  TOS at 4 hrs for episode 12 (n=13) | 76.92 (43.853)
  TOS at 4 hrs for episode 13 (n=12) | 64.93 (46.854)

3. Secondary Outcome: Time to Significant Improvement
Description: Time to significant improvement in overall response based on the period from 15 minutes after dosing through 4 hrs post dosing. Significant improvement was defined as a response of "a lot better or resolved" in the overall response assessment.
Time Frame: 15 min - 4 hrs post dose after every episode
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: estimated time in minutes
Arm/Group | DX-88 (Ecallantide)
Number analyzed (Participants) | 145
estimated time in minutes
  time to improvement in min. for episode 1 (n=145) | 225.2 [165.4 to 228.2]
  time to improvement in min. for episode 2 (n=102) | 194.5 [165.2 to 227.5]
  time to improvement in min. for episode 3 (n=77) | 225.4 [225.1 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.
  time to improvement in min. for episode 4 (n=56) | 198.1 [165.4 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.
  time to improvement in min. for episode 5 (n=41) | 240.0 [165.3 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.
  time to improvement in min. for episode 6 (n=33) | 225.2 [137.0 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.
  time to improvement in min. for episode 7 (n=27) | NA [195.3 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.
  time to improvement in min. for episode 8 (n=23) | 210.5 [135.3 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.
  time to improvement in min. for episode 9 (n=23) | 169.3 [135.4 to 240.0]
  time to improvement in min. for episode 10 (n=17) | 170.5 [165.1 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.
  time to improvement in min. for episode 11 (n=16) | 226.5 [145.7 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.
  time to improvement in min. for episode 12 (n=15) | 177.2 [113.8 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.
  time to improvement in min. for episode 13 (n=13) | 195.2 [135.1 to NA] — N/A: significant improvement in overall response was not reached within 4 hours.

ADVERSE EVENTS:
Time Frame: pre-dose to 28 days (+/-2 days) post dose
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 27/147
Other Adverse Events (participants affected / at risk) | 102/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=147)
hereditary angioedema (Congenital, familial and genetic disorders) | 17 (17)
hypersensitivity (Immune system disorders) | 1 (1)
anaphylactic reaction (Immune system disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 4 (4)
cholecystitis (Hepatobiliary disorders) | 1 (1)
otitis externa (Infections and infestations) | 1 (1)
cellulitis staphyloccal (Infections and infestations) | 1 (1)
contusion (Injury, poisoning and procedural complications) | 1 (1)
transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
liver function test abnormal (Investigations) | 1 (1)
white blood cell count increased (Investigations) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1)
laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
erythema (Skin and subcutaneous tissue disorders) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
homicide (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=147)
hereditary angioedema (Congenital, familial and genetic disorders) | 25 (25)
nausea (Gastrointestinal disorders) | 19 (19)
headache (Nervous system disorders) | 16 (16)
abdominal pain (Gastrointestinal disorders) | 12 (12)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 11 (11)
vomiting (Gastrointestinal disorders) | 10 (10)
diarrhoea (Gastrointestinal disorders) | 9 (9)
anxiety (Psychiatric disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Dyax agreements vary, but Dyax will not prohibit any investigator from publishing. Dyax reviews publications prior to public release and can request deferral by up to 60 days beyond the proposed publication date if necessary to preserve its intellectual property. Dyax can request changes to publications to remove non-study-related confidential information. Dyax can also request deferral of single-center publications until after disclosure of the clinical trial's primary publication.